CLINICAL TRIAL: NCT03461211
Title: Multicenter, Safety and Efficacy, Open-Label Extension Study Evaluating Teprotumumab (HZN-001) Treatment in Subjects With Thyroid Eye Disease
Brief Title: Treatment of Graves' Orbitopathy to Reduce Proptosis With Teprotumumab Infusions in an Open-Label Clinical Extension Study
Acronym: OPTIC-X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-TEP-302; 2017-002713-58 (EudraCT Number)
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teprotumumab (Experimental): Eight infusions of teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
  Interventions: Biological: Teprotumumab

INTERVENTIONS:
Biological: Teprotumumab — Teprotumumab is a fully human anti-IGF-1R mAb. Teprotumumab will be provided in single-dose 20 mL glass vials as a freeze-dried powder. Each vial of teprotumumab must be reconstituted with 10 mL of water for injection. Reconstituted teprotumumab solution must be further diluted in 0.9% (w/v) sodium chloride (NaCl) solution prior to administration. Teprotumumab will be administered in 100 mL or 250 mL infusion bags (100 mL infusion bags for doses up to 1800 mg and 250 mL infusion bags for doses > 1800 mg).
  Other Names: HZN-001

SUMMARY:
The overall objective is to evaluate the safety and efficacy of teprotumumab in the treatment of thyroid eye disease (TED) in participants who participated in the lead-in study HZNP-TEP-301 (NCT03298867; OPTIC) and who were either proptosis non-responders at Week 24 of HZNP-TEP-301 or were proptosis responders at Week 24 but met the criteria for re-treatment due to relapse during the Follow-Up Period of HZNP-TEP-301.

DETAILED DESCRIPTION:
This is a multi-center, open-label extension study of HZNP-TEP-301 (NCT03298867) examining the safety and efficacy of teprotumumab in the treatment of TED in adult participants. Participants who complete the 24-week double-masked Treatment Period in Study HZNP-TEP-301 and are proptosis non-responders or are proptosis responders at Week 24 but meet the criteria for re-treatment due to relapse during the Follow-Up Period of HZNP-TEP-301 will be eligible for enrollment.

All participants who choose to participate will receive 8 infusions of teprotumumab (10 mg/kg for the first infusion followed by 20 mg/kg for the remaining 7 infusions) in an open-label fashion. The Baseline (Day 1) Visit of this extension study will occur within 14 days after the final visit of Study HZNP-TEP-301 (Week 24 for proptosis non-responders and up to Week 72 for participants who relapse). During the open-label Treatment Period, study drug infusions are scheduled for Day 1 (Baseline), and Weeks 3, 6, 9, 12, 15, 18, and 21, (with the final visit at Week 24). After completion of the Treatment Period, subjects who were proptosis non-responders in Study HZNP-TEP-301 will enter a 24-week Follow-Up Period during which study drug will not be administered and clinic visits are scheduled for 1, 3, and 6 months (Visits Month 7, 9, and 12) after the Week 24 visit. Subjects will be contacted 6 and 12 months later by phone or email to enquire if any treatment for TED had been received since the last study contact.

Participants who relapse during the Follow-Up Period of HZNP-TEP-301 and choose to enter this extension study will not participate in the Follow-Up Period of this study but will be contacted by phone or email 6 and 12 months after the Week 24 visit.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Completed the 24-week double-masked Treatment Period in Study HZNP-TEP-301 (NCT03298867).
* Proptosis non-responder (< 2 mm reduction in proptosis in the study eye) at Week 24 of Study HZNP-TEP-301 OR proptosis responder at Week 24 who relapses during the Follow-Up Period of Study HZNP-TEP-301.
* Participant must be euthyroid with the baseline disease under control, or have mild hypo- or hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine [FT3] levels < 50% above or below the normal limits) at the most recent clinic visit. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of the clinical trial.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN) or serum creatinine <1.5 times the upper limit of normal (ULN; according to age) at the most recent clinic visit.
* Diabetic participants must have well-controlled disease (defined as hemoglobin A1C [HbA1c] < 9.0% at most recent clinic visit).
* Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the course of the study.
* Women of childbearing potential must have a negative urine pregnancy test at Baseline/Day 1. Participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial and continue for 180 days after the last dose of study drug. One of the 2 forms of contraception is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be in use for at least one full cycle prior to Baseline. Highly effective contraceptive methods (with a failure rate less than 1% per year), when used consistently and correctly, includes implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner.
* Male participants must be surgically sterile or, if sexually active with a female partner of childbearing potential, must agree to use a barrier contraceptive method from Baseline through 180 days after the last dose of study drug.
* Participant is willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.
* Has not received any treatment for TED since Week 24 of the of the HZNP-TEP-301 study.

Exclusion Criteria:

* Participants will be ineligible if, in the opinion of the Investigator, they are unlikely to comply with the study protocol or have a concomitant disease or condition that could interfere with the conduct of the study or potentially put the participant at unacceptable risk.
* The exclusion criteria (except those related to screening) of protocol HZNP-TEP-301(NCT03298867) also apply to this open-label extension study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (8):
  - Macro, Llc, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Kellogg Eye Center at University of Michigan, Ann Arbor, Michigan
  - Casey Eye Institute at Oregon Health and Science, Portland, Oregon
  - Hamilton Eye Institute at University of Tennessee Health, Memphis, Tennessee
  - Eye Wellness Center, Houston, Texas
  - Medical College of Wisconsin, The Eye Institute, Milwaukee, Wisconsin
- Germany (2):
  - University Hospital Essen, Department of Ophthalmology, Essen
  - Johannes Gutenberg University Medical Center, Mainz
- Italy (3):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore, Milan
  - University of Pisa, Department of Clinical and Experimental Medicine, Pisa
  - Azienda Ospedaliero Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Xin Y, Xu F, Gao Y, Bhatt N, Chamberlain J, Sile S, Hammel S, Holt RJ, Ramanathan S. Pharmacokinetics and Exposure-Response Relationship of Teprotumumab, an Insulin-Like Growth Factor-1 Receptor-Blocking Antibody, in Thyroid Eye Disease. Clin Pharmacokinet. 2021 Aug;60(8):1029-1040. doi: 10.1007/s40262-021-01003-3. Epub 2021 Mar 26. PMID 33768488
- See also: Related Info — http://www.TEPEZZA.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible for enrollment in this study (OPTIC-X) if they completed the 24-week double-masked Treatment Period in Study HZNP-TEP-301 (NCT03298867; OPTIC) and were proptosis non-responders or were proptosis responders at Week 24 but met the criteria for re-treatment due to relapse during the Follow-Up Period of HZNP-TEP-301.
Pre-assignment Details: The Baseline (Day 1) Visit of this extension study occurred within 14 days after the final visit of Study HZNP-TEP-301, which was Week 24 for proptosis non-responders and up to Week 72 for participants who relapsed.
  The study treatment previously administered in HZNP-TEP-301 (teprotumumab or placebo) remained masked throughout this extension study.
Groups:
- Teprotumumab (OPTIC Placebo): Participants who received placebo in OPTIC received 8 infusions of open-label teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Teprotumumab (OPTIC Teprotumumab): Participants who received teprotumumab in OPTIC received 8 infusions of open-label teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
Period: Overall Study
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Started | 37 | 14
Proptosis Non-Responders in OPTIC | 36 | 5
Relapsed During Follow-Up Period of OPTIC | 1 | 9
Completed | 36 | 12
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Teprotumumab (OPTIC Placebo): Participants who received placebo in OPTIC received 8 infusions of teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Teprotumumab (OPTIC Teprotumumab): Participants who received teprotumumab in OPTIC received 8 infusions of teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Total: Total of all reporting groups
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab) | Total
Number analyzed (Participants) | 37 | 14 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (13.49) | 56.1 (11.52) | 50.6 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 11 | 38
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 36 | 14 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 1 | 1 | 2
  White | 33 | 11 | 44
  Other, Not Specified | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 2 mm Reduction From Baseline in the Study Eye Without Deterioration of Proptosis in the Fellow Eye at Week 24
Description: Proptosis responders were defined as participants with a ≥ 2 mm reduction from study baseline in proptosis in the study eye, without deterioration (≥ 2 mm increase) of proptosis in the fellow eye at Week 24. Participants missing Week 24 values were considered non-responders, aside from those with missing data related to the COVID-19 pandemic.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat Population: all participants enrolled in the study. Participants missing Week 24 values were considered non-responders, aside from those with missing data related to the COVID-19 pandemic. One participant in the Teprotumumab (OPTIC Teprotumumab) arm was excluded from all Week 24 summaries due to COVID-19 (visit delayed).
Measure: Number; unit: percentage of participants
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Number analyzed (Participants) | 37 | 13
percentage of participants | 89.2 | 53.8

2. Secondary Outcome: Percentage of Participants With a European Group on Graves' Ophthalmopathy (EUGOGO) Amended Clinical Activity Score (CAS) Total Score of 0 or 1 in the Study Eye at Week 24
Description: CAS responders were defined as participants with a reduction to a CAS of 0 or 1 (no or minimal inflammatory symptoms) as a categorical response variable at Week 24.
  The 7-item CAS assigns 1 point for each of the following items present in the study eye: spontaneous orbital pain; gaze evoked orbital pain; eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/Graves' ophthalmopathy (TED/GO); eyelid erythema; conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness); chemosis; inflammation of caruncle or plica. The sum of these points is the total score (0 to 7), with higher scores indicating worse symptoms.
Time Frame: Week 24
Population: Intent-to-Treat Population: all participants enrolled in the study. Participants with CAS > 1 at Study Baseline. Per the statistical analysis plan, participants missing Week 24 values were considered non-responders, aside from those with missing data related to the COVID-19 pandemic. One participant in the Teprotumumab (OPTIC Teprotumumab) arm was excluded from all Week 24 summaries due to COVID-19 (visit delayed).
Measure: Number; unit: percentage of participants
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Number analyzed (Participants) | 32 | 11
percentage of participants | 65.6 | 36.4

3. Secondary Outcome: Change in Proptosis From Baseline to Week 24
Description: Mean change from study baseline to Week 24 in proptosis measurement (mm) in the study eye at Week 24.
Time Frame: Study Baseline, Week 24
Population: Intent-to-Treat Population: all participants enrolled in the study. Participants with both baseline and Week 24 measurements. One participant in the Teprotumumab (OPTIC Teprotumumab) arm was excluded from all Week 24 summaries due to COVID-19 (visit delayed).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Number analyzed (Participants) | 36 | 11
mm | -3.47 (1.732) | -1.77 (1.126)

4. Secondary Outcome: Percentage of Participants Who Were Diplopia Responders at Week 24
Description: Diplopia responders were defined as participants with 1 grade or greater reduction in diplopia score in the study eye without worsening by at least 1 grade in the fellow eye at Week 24.
  The subjective diplopia score (0=no diplopia; 1=intermittent, i.e. diplopia in primary position of gaze, when tired or when first awakening; 2=inconstant, i.e. diplopia at extremes of gaze; 3=constant, i.e. continuous diplopia in primary or reading position) was recorded for each eye. A participant was considered to have diplopia if a score > 0 is observed in the study eye at study baseline.
Time Frame: Week 24
Population: Intent-to-Treat Population: all participants enrolled in the study. Participants with diplopia at Study Baseline. Per the statistical analysis plan, participants missing Week 24 values were considered non-responders, aside from those with missing data related to the COVID-19 pandemic. One participant in the Teprotumumab (OPTIC Teprotumumab) arm was excluded from all Week 24 summaries due to COVID-19 (visit delayed).
Measure: Number; unit: percentage of participants
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Number analyzed (Participants) | 23 | 4
percentage of participants | 60.9 | 75.0

5. Secondary Outcome: Mean Change From Baseline to Week 24 in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire Overall Score
Description: The GO-QoL is a 16-item self-administered questionnaire divided into 2 subsets and used to assess the perceived effects of TED by the participants on (i) their daily physical activity as it relates to visual function, and (ii) psychosocial functioning. The sum of the scores from each set of 8 questions was calculated and transformed to a scale from 0 (worst) to 100 (best) - one for visual function (VF), one for appearance (A) and one for the overall combined (VF + A) score. Scores were transformed as follows: Transformed score = [(sum of each score - number of completed items) / (2 * number of completed items)] * 100. The "overall combined (VF + A) score" is also 0 to 100, with higher scores indicating a better outcome.
Time Frame: Study Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teprotumumab (OPTIC Placebo) | Teprotumumab (OPTIC Teprotumumab)
Number analyzed (Participants) | 36 | 11
score on a scale | 13.39 (17.890) | 14.73 (11.777)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious Adverse Events (AEs): from informed consent through 30 days after study discontinuation. Mean days on study was 332.9 and 218.8 for Teprotumumab (OPTIC Placebo) and Teprotumumab (OPTIC Teprotumumab) arms, respectively.
Description: Non-serious AEs: from first dose of study drug through last dose of study drug + 3 weeks (Treatment Period; mean 168.1 and 170.9 days for Placebo and Teprotumumab arms, respectively) or from Week 24 up to Week 48 in the Follow-Up Period (mean 170.1 and 165.0 days for Teprotumumab (OPTIC Placebo) and Teprotumumab (OPTIC Teprotumumab) arms, respectively).
Groups:
- Treatment Period: Teprotumumab (OPTIC Placebo): Participants who received placebo in OPTIC received 8 infusions of teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Treatment Period: Teprotumumab (OPTIC Teprotumumab): Participants who received teprotumumab in OPTIC received 8 infusions of teprotumumab every 3 weeks (q3W) for a total of 21 weeks: teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Follow-Up Period: No Treatment (OPTIC Placebo): Participants who received placebo in OPTIC and were proptosis non-responders. Participants received 8 infusions of teprotumumab q3W for a total of 21 weeks in OPTIC-X and entered a 24-week Follow-up Period; no trial drug was administered.
- Follow-Up Period: No Treatment (OPTIC Teprotumumab): Participants who received teprotumumab in OPTIC and were proptosis non-responders. Participants received 8 infusions of teprotumumab q3W for a total of 21 weeks in OPTIC-X and entered a 24-week Follow-up Period; no trial drug was administered.
Arm/Group | Treatment Period: Teprotumumab (OPTIC Placebo) | Treatment Period: Teprotumumab (OPTIC Teprotumumab) | Follow-Up Period: No Treatment (OPTIC Placebo) | Follow-Up Period: No Treatment (OPTIC Teprotumumab)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/14 | 0/36 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/14 | 0/36 | 0/4
Other Adverse Events (participants affected / at risk) | 32/37 | 11/14 | 16/36 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Teprotumumab (OPTIC Placebo) (N=37) | Treatment Period: Teprotumumab (OPTIC Teprotumumab) (N=14) | Follow-Up Period: No Treatment (OPTIC Placebo) (N=36) | Follow-Up Period: No Treatment (OPTIC Teprotumumab) (N=4)
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Teprotumumab (OPTIC Placebo) (N=37) | Treatment Period: Teprotumumab (OPTIC Teprotumumab) (N=14) | Follow-Up Period: No Treatment (OPTIC Placebo) (N=36) | Follow-Up Period: No Treatment (OPTIC Teprotumumab) (N=4)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Autophony (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 3 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 2 | 1 | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Lenticular Opacities (Eye disorders) | 1 | 0 | 0 | 0
Ocular Discomfort (Eye disorders) | 1 | 0 | 0 | 0
Punctate Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gingival Recession (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Noninfective Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue Ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0
Sinusitis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural Headache (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0
Weight Increased (Investigations) | 1 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 18 | 4 | 3 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Haemangioma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Balance Disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0
Visual Field Defect (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0
Tension (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Jugular Vein Distension (Vascular disorders) | 1 | 0 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Pupillary Reflex Impaired (Eye disorders) | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Post Procedural Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
White Matter Lesion (Nervous system disorders) | 0 | 0 | 0 | 1
Diffuse Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT03461211/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03461211/SAP_001.pdf